CLINICAL TRIAL: NCT00528879
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Phase III Study of BMS-512148 (Dapagliflozin) in Patients With Type 2 Diabetes Who Are Not Well Controlled on Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-014 LT; MB102-014 (Other: Other Study ID Numbers:)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Metformin; Hypoglycemic Agents; Pharmacologic Actions; Physiological Effects of Drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + Metformin (Placebo Comparator): Participants received dapagliflozin-matching placebo once daily plus open-label metformin ≥1500 mg per day for up to 102 weeks
  Interventions: Drug: Placebo; Drug: Metformin
- Dapagliflozin, 2.5 mg + Metformin (Experimental): Participants received dapagliflozin, 2.5 mg, once daily plus open-label metformin ≥1500 mg per day for up to 102 weeks
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Dapagliflozin, 5 mg + Metformin (Experimental): Participants received dapagliflozin, 5 mg, once daily plus open-label metformin ≥1500 mg per day for up to 102 weeks
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Dapagliflozin, 10 mg + Metformin (Experimental): Participants received dapagliflozin, 10 mg, once daily plus open-label metformin ≥1500 mg per day for up to 102 weeks
  Interventions: Drug: Dapagliflozin; Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets administered orally as a 2.5-, 5-, or 10-mg dose once daily for up to 102 weeks
  Other Names: BMS-512148
  Arms: Dapagliflozin, 10 mg + Metformin; Dapagliflozin, 2.5 mg + Metformin; Dapagliflozin, 5 mg + Metformin
Drug: Placebo — Dapagliflozin-matching placebo administered as tablets orally once daily for up to 102 weeks
  Arms: Dapagliflozin, 10 mg + Metformin; Placebo + Metformin
Drug: Metformin — Open-label metformin administered as ≥1500 mg per day for up to 102 weeks

SUMMARY:
The purpose of this clinical research study is to learn whether dapagliflozin can help reduce blood sugar levels in participants with Type 2 diabetes that is not well controlled on metformin alone. The safety of this treatment will also be studied.

ELIGIBILITY:
Key Inclusion Criteria

* Males and females, 18 to 77 years old, with type 2 diabetes and inadequate glycemic control
* Participants who have been receiving metformin at a total daily dose ≥1500 mg per day for at least 8 weeks
* C-peptide ≥1.0 ng/mL
* Body mass index ≤45.0 kg/m^2
* Serum creatinine level <1.50 mg/dL for men or <1.40 mg/dL for women.

Key Exclusion Criteria

* Aspartate aminotransferase and/or alanine aminotransferase level >3.0 times the upper limit of normal
* Serum total bilirubin level >2 mg/dL
* Creatinine kinase level >3 times upper limit of normal
* Symptoms of severely uncontrolled diabetes
* Serum creatinine level ≥1.50 mg/dL for men or ≥1.40 mg/dL for women
* Currently unstable or serious cardiovascular, renal, hepatic, hematologic, oncologic, endocrine, psychiatric, or rheumatic diseases

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (67):
- United States (28):
  - Clinical Research Advantage / Desert Clinical Res, Llc, Tempe, Arizona
  - Medical Group Of Encino, Encino, California
  - Valley Research, Fresno, California
  - Randall Shue, D.O., Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Ritchken & First M.D.'S, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Raikhel, Marina, Torrance, California
  - Express Care Clinical Res, Colorado Springs, Colorado
  - Denver Internal Medicine, Denver, Colorado
  - New West Physicians, Golden, Colorado
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Family Care Associates Of Nw Florida, Chipley, Florida
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Woodlake Research, Chesterfield, Missouri
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - Diabetes & Endocrinology Consultants, Pc, Morehead City, North Carolina
  - Newark Physician Associates, Newark, Ohio
  - Integris Family Care S. Penn, Oklahoma City, Oklahoma
  - Cumberland Valley Endocrinology Center, Llc, Carlisle, Pennsylvania
  - Banksville Medical Pc, Pittsburgh, Pennsylvania
  - Palmetto Clinical Research, Summerville, South Carolina
  - Southeastern Research Assoc, Taylors, South Carolina
  - Texas Center For Drug Development, P.A., Houston, Texas
  - Diabetes & Glandular Disease Research Associates, Inc., San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Optimum Clinical Research, Salt Lake City, Utah
  - Office Of Dr. Gray, Spokane, Washington
- Argentina (8):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Auton., Buenos Aires
  - Local Institution, Ciudad Auton, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Zárate, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Villa Carlos Paz, Córdoba Province
- Brazil (7):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Itajubá, Minas Gerais
  - Local Institution, Belém, Pará
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Caxias do Sul, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Marília, São Paulo
- Canada (16):
  - Local Institution, Calgary, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Sarnia, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, L'Ancienne-Lorette, Quebec
  - Local Institution, Mirabel, Quebec
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (8):
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Guadalajara, Mexico City
  - Local Institution, Zapopan, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrrey, Nuevo León
  - Local Institution, Tampico, Tamaulipas

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Shah M, Stolbov L, Yakovleva T, Tang W, Sokolov V, Penland RC, Boulton D, Parkinson J. A model-based approach to investigating the relationship between glucose-insulin dynamics and dapagliflozin treatment effect in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Apr;23(4):991-1000. doi: 10.1111/dom.14305. Epub 2021 Jan 25. PMID 33368935
- [Derived] Bailey CJ, Del Prato S, Wei C, Reyner D, Saraiva G. Durability of glycaemic control with dapagliflozin, an SGLT2 inhibitor, compared with saxagliptin, a DPP4 inhibitor, in patients with inadequately controlled type 2 diabetes. Diabetes Obes Metab. 2019 Nov;21(11):2564-2569. doi: 10.1111/dom.13841. Epub 2019 Aug 26. PMID 31364269
- [Derived] Mellander A, Billger M, Johnsson E, Traff AK, Yoshida S, Johnsson K. Hypersensitivity Events, Including Potentially Hypersensitivity-Related Skin Events, with Dapagliflozin in Patients with Type 2 Diabetes Mellitus: A Pooled Analysis. Clin Drug Investig. 2016 Nov;36(11):925-933. doi: 10.1007/s40261-016-0438-3. PMID 27461213
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- [Derived] Bailey CJ, Gross JL, Hennicken D, Iqbal N, Mansfield TA, List JF. Dapagliflozin add-on to metformin in type 2 diabetes inadequately controlled with metformin: a randomized, double-blind, placebo-controlled 102-week trial. BMC Med. 2013 Feb 20;11:43. doi: 10.1186/1741-7015-11-43. PMID 23425012
- [Derived] Bailey CJ, Gross JL, Pieters A, Bastien A, List JF. Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with metformin: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Jun 26;375(9733):2223-33. doi: 10.1016/S0140-6736(10)60407-2. PMID 20609968

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 915 participants enrolled, 562 completed a qualification period. Of these 562 participants, 546 were randomized and received treatment and 16 were excluded due to adverse events (1), no longer meeting study criteria (7), poor compliance or noncompliance (3), withdrawn consent (4), and lost to follow-up (1).
Period: Short-term Period (Day 1 to Week 24)
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Started | 137 | 137 | 137 | 135
Completed the Period | 119 | 121 | 122 | 121
Completed | 115 (Completed=entered Long-term Period) | 120 (Completed=entered Long-term Period) | 122 (Completed=entered Long-term Period) | 119 (Completed=entered Long-term Period)
Not Completed | 22 | 17 | 15 | 16
Not completed — Lack of Efficacy | 3 | 0 | 1 | 0
Not completed — Adverse Event | 4 | 4 | 2 | 4
Not completed — Withdrawal by Subject | 7 | 5 | 5 | 3
Not completed — Lost to Follow-up | 5 | 4 | 4 | 5
Not completed — Poor compliance/noncompliance | 0 | 0 | 2 | 0
Not completed — No longer meets study criteria | 2 | 3 | 0 | 2
Not completed — Administrative reason by author | 1 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 1
Period: Long-term Period (Weeks 24 to 102)
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Started | 115 | 120 | 122 | 119
Completed | 73 | 82 | 89 | 95
Not Completed | 42 | 38 | 33 | 24
Not completed — Lack of Efficacy | 27 | 16 | 17 | 9
Not completed — Adverse Event | 5 | 4 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 6 | 8 | 4
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 5 | 3 | 7
Not completed — Poor compliance/noncompliance | 0 | 5 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — No longer meets study criteria | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin | Total
Number analyzed (Participants) | 137 | 137 | 137 | 135 | 546
Age, Continuous [Mean (Full Range); unit: Years] | 53.7 [30 to 74] | 55.0 [30 to 76] | 54.3 [33 to 75] | 52.7 [29 to 76] | 53.9 [29 to 76]
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 114 | 116 | 119 | 118 | 467
  65 to younger than 75 years | 23 | 19 | 17 | 16 | 75
  75 years and older | 0 | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 67 | 68 | 58 | 254
  Male | 76 | 70 | 69 | 77 | 292
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 124 | 117 | 118 | 121 | 480
  Black/African American | 2 | 5 | 6 | 4 | 17
  Asian | 3 | 3 | 4 | 1 | 11
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  American Indian/Alaskan Native | 1 | 2 | 2 | 4 | 9
  Other | 7 | 10 | 6 | 5 | 28
Female Age [Number; unit: Participants]
  50 Years and younger | 25 | 18 | 22 | 22 | 87
  Older than 50 years | 36 | 49 | 46 | 36 | 167
Body Mass Index [Number; unit: Participants]
  <25 kg/m^2 | 9 | 4 | 12 | 12 | 37
  ≥25 kg/m^2 | 128 | 133 | 125 | 123 | 509
  ≥27 kg/m^2 | 115 | 120 | 111 | 106 | 452
  ≥30 kg/m^2 | 79 | 77 | 81 | 75 | 312

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 134 | 135 | 133 | 132
Percent | -0.30 (0.0718) | -0.67 (0.0715) | -0.70 (0.0722) | -0.84 (0.0724)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; p = 0.0002, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Mean Difference (Final Values) = -0.38, Standard Error of Mean 0.1014
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Mean Difference (Final Values) = -0.41, Standard Error of Mean 0.1016
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Mean Difference (Final Values) = -0.54, Standard Error of Mean 0.1021

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Data after rescue medication was excluded from this analysis. Fasting plasma glucose was measured as milligrams per deciliter (mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and who had nonmissing fasting plasma glucose values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 136 | 137 | 136 | 132
mg/dL | -6.0 (2.673) | -17.8 (2.663) | -21.5 (2.679) | -23.5 (2.721)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; p < 0.0019, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -11.8, Standard Error of Mean 3.774
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -15.5, Standard Error of Mean 3.781
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -17.5, Standard Error of Mean 3.819

3. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing total body weights at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 136 | 137 | 137 | 133
Kilograms | -0.89 (0.2368) | -2.21 (0.2357) | -3.04 (0.2358) | -2.86 (0.2392)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -1.32, Standard Error of Mean 0.3344
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -2.16, Standard Error of Mean 0.3344
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -1.97, Standard Error of Mean 0.3365

4. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Percent adjusted for baseline HbA1c. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and were not missing baseline and Week 24 (LOCF) values
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 134 | 135 | 133 | 132
Percentage of participants | 25.9 | 33.0 | 37.5 | 40.6
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; p = 0.1775, Modified logistic regression — Statistically significant according to hierarchical testing procedure (p<0.05); Median Difference (Final Values) = 7.1
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p = 0.0275, Modified logistic regression — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = 11.7
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p = 0.0062, Modified logistic regression — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = 14.7

5. Secondary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) in Participants With Baseline HbA1c ≥9.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. HbA1c was measured as percent of hemoglobin by a central laboratory. The population included those randomized participants who received treatment and had a baseline HbA1c > 9.0%. Data after rescue medication were excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication, who had baseline HbA1c ≥9.0%, and who had nonmissing HbA1c values at Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 22 | 17 | 34 | 18
Percent | -0.53 (0.2345) | -1.21 (0.2660) | -1.37 (0.1875) | -1.32 (0.2595)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; ANCOVA — Sequential testing procedures were used, and no test was performed for this comparison due to the fact that the previous comparison was not significant; Mean Difference (Final Values) = -0.68, Standard Error of Mean 0.3515
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p = 0.0068, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -0.84, Standard Error of Mean 0.3022
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p = 0.0290, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -0.78, Standard Error of Mean 0.3535

6. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight at Week 24 in Participants With Baseline Body Mass Index (BMI) ≥27 kg/m^2 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined.) Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in Periods and on Day 1 and Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication, who had baseline BMI ≥27 kg/m^2, and who had nonmissing total body weight measurements at Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 114 | 120 | 111 | 108
Kilograms | -1.01 (0.2630) | -2.39 (0.2564) | -3.21 (0.2661) | -3.09 (0.2737)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.38, Standard Error of Mean 0.3681
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -2.19, Standard Error of Mean 0.3745
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -2.08, Standard Error of Mean 0.3791

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Hypoglycemia Events, Related AEs, Death as Outcome, Serious AEs (SAEs), Related SAEs, SAEs Leading to Discontinuation, AEs Leading to Discontinuation, and Hypoglycemia Events Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or missing relationship to study drug. Events captured from baseline to last dose plus 4 days for AEs and plus 30 days for SAEs during the double-blind 12-week period. Data after rescue included.
Time Frame: From Baseline to end of Long-term Period (Week 102)
Population: All randomized participants who received at least 1 dose of blinded study medication
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 137 | 137 | 137 | 135
Participants
  At least 1 AE | 111 | 111 | 111 | 111
  At least 1 hypoglycemia event | 8 | 5 | 7 | 7
  At least 1 related AE | 28 | 36 | 33 | 45
  Deaths | 1 | 2 | 0 | 0
  At least 1 SAE | 14 | 15 | 9 | 14
  At least 1 related SAE | 3 | 0 | 2 | 1
  SAEs leading to discontinuation | 6 | 3 | 1 | 2
  AEs leading to discontinuation | 9 | 7 | 5 | 6
  Hypoglycemia events leading to discontinuation | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Laboratory Abnormality
Description: BUN=blood urea nitrogen; preRX=pretreatment; ULN=upper limit of normal; AST=aspartate aminotransferase; ALT=alanine aminotransferase; ALP=alkaline phosphatase. Phosphorus, inorganic (low): ages 17-65 years, ≤1.8 mg/dL; ages≥66 years, ≤2.1 mg/dL. Phosphorus, inorganic (high): ages 17-65 years, ≥5.6 mg/dL; ages≥66 years, ≥5.6 mg/dL. Phosphorus, inorganic (low) ≤1.8 mg/dL if age 17-65 or ≤2.1 mg/dL if age ≥66. Calcium, total (high): ≥1 mg/dL from ULN and ≥0.5 mg/dL from preRx value.
Time Frame: Day 1 to Week 102
Population: All randomized participants who received at least 1 dose of study medication and who had nonmissing laboratory values at baseline and Week 102.
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 136 | 137 | 136 | 132
Participants
  Hematocrit >55% | 1 | 2 | 2 | 3
  Hemoglobin >18 g/dL | 1 | 4 | 1 | 5
  BUN ≥60 mg/d or Urea>21.4 mmol/L | 0 | 0 | 0 | 1
  Creatinine ≥1.5 preRX creatinine | 2 | 3 | 4 | 2
  Creatinine ≥2.5 mg/dL | 0 | 0 | 1 | 0
  Glucose >350 mg/dL | 2 | 0 | 0 | 1
  Creatine kinase >5*ULN | 2 | 2 | 3 | 3
  Creatine kinase >10*ULN | 1 | 0 | 2 | 1
  Calcium, total <7.5 mg/dL | 4 | 1 | 2 | 0
  Calcium, total (high) | 2 | 0 | 0 | 0
  Potassium, serum ≥6 MEQ/L | 6 | 3 | 3 | 2
  Magnesium, serum <1 mEq/L | 1 | 0 | 0 | 1
  Sodium, serum <130 mEq/L | 1 | 0 | 3 | 0
  Sodium, serum >150 mEq/L | 0 | 0 | 1 | 0
  Phosphorus, inorganic (high) | 1 | 1 | 2 | 5
  Phosphorus, inorganic (low) | 1 | 0 | 0 | 0
  Albumin/creatinine ratio >1800 mg/g | 2 | 0 | 3 | 1
  AST elevation 3*ULN | 0 | 0 | 3 | 2
  ALT elevation 3*ULN | 1 | 3 | 2 | 2
  ALT elevation 5*ULN | 0 | 0 | 1 | 0
  Total bilirubin elevation >1.5*ULN | 2 | 1 | 1 | 4
  Total bilirubin elevation >2*ULN | 0 | 0 | 0 | 1
  ALP elevation >1.5*ULN | 5 | 5 | 0 | 2

9. Other Pre Specified Outcome: Number of Participants With Changes in Baseline in Electrocardiogram Findings at Week 102 (Last Observation Carried Forward [LOCF])
Description: 12-Lead electrocardiograms (ECGs) were performed at entry into lead-in period Day -7 visit and Week 24/dnd of treatment visit (LOCF) on participants who were supine. ECGs were assessed by the investigator. Baseline was Day -7 for this parameter. Data after rescue included.The Week 102 value is the last observation, regardless of rescue prior to Week 102 if no Week 102 measurement was available.
Time Frame: Baseline to Week 102
Population: All randomized participants who received at least 1 dose of study medication and who had nonmissing baseline and Week 102 (LOCF) values
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 137 | 137 | 137 | 135
Participants
  Baseline normal/Week 102 normal | 74 | 80 | 79 | 82
  Baseline normal/Week 102 abnormal | 7 | 14 | 9 | 8
  Baseline normal/Week 102 not reported | 9 | 6 | 5 | 9
  Baseline abnormal/Week 102 normal | 17 | 11 | 20 | 10
  Baseline abnormal/Week 102 abnormal | 26 | 24 | 20 | 25
  Baseline abnormal/Week 102 not reported | 3 | 2 | 3 | 1
  Baseline not reported/Week 102 normal | 1 | 0 | 1 | 0
  Baseline not reportedl/Week 102 abnormal | 0 | 0 | 0 | 0
  Baseline not reported/Week 102 not reported | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Mean Changes From Baseline in Seated Systolic Blood Pressure
Description: Blood pressure values were obtained after the participant was seated quietly for 5 minutes; at least 8 hours after the last ingestion of caffeine, alcohol, or nicotine; and in the same arm (right or left) consistently through out the study. Data after rescue were also included. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 102
Population: All randomized participants who received study medication. n=the number of participants not missing baseline and Week t values.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 137 | 137 | 137 | 135
mm Hg
  Week 12 (n=125, 129, 129, 126) | -0.1 (1.216) | -1.6 (1.380) | -4.0 (1.206) | -3.0 (1.230)
  Week 24 (n=119, 119, 122, 122) | -0.2 (1.229) | -2.1 (1.126) | -4.3 (1.270) | -5.1 (1.329)
  Week 50 (n=105, 116, 111, 113) | 1.0 (1.440) | -0.1 (1.281) | -2.1 (1.314) | -1.9 (1.472)
  Week 102 (n=72, 78, 88, 94) | 1.5 (1.610) | 0.7 (1.825) | -1.1 (1.412) | -0.3 (1.544)

11. Other Pre Specified Outcome: Mean Changes From Baseline in Seated Diastolic Blood Pressure
Description: as for outcome 10
Time Frame: From Baseline to Week 102
Population: as for outcome 10
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 137 | 137 | 137 | 135
mm Hg
  Week 12 (n=125, 129, 129, 126) | -0.9 (0.763) | -1.3 (0.794) | -2.3 (0.714) | -1.0 (0.758)
  Week 24 (n=119, 119, 122, 122) | -0.1 (0.744) | -1.8 (0.863) | -2.5 (0.769) | -1.8 (0.842)
  Week 50 (n=105, 116, 111, 113) | 0.1 (0.861) | -0.2 (0.714) | -2.4 (0.840) | -1.2 (0.921)
  Week 102 (n=72, 78, 88, 94) | -1.0 (0.929) | -0.1 (0.914) | -1.5 (0.861) | -1.2 (1.041)

12. Other Pre Specified Outcome: Number of Participants With Orthostatic Hypotension
Description: Orthostatic hypotension was defined as a decrease from supine to standing blood pressure of >20 mm Hg in systolic blood pressure or >10 mm Hg in diastolic blood pressure.
Time Frame: From Baseline to Week 102
Population: All randomized participants who received treatment; n=the number of participants who were not missing blood pressure measurements.
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 137 | 137 | 137 | 135
Participants
  Baseline (n=121, 127, 124, 126) | 3 | 4 | 4 | 4
  Week 1 (n=126, 121, 119, 114) | 28 | 26 | 21 | 19
  Week 12 (n=123, 128, 127, 125) | 6 | 8 | 4 | 5
  Week 24 (n=116, 114, 118, 121) | 10 | 6 | 5 | 3
  Week 50 (n=103, 115, 109,112) | 10 | 6 | 7 | 6
  Week 102 (n=71, 76, 87, 94) | 1 | 1 | 1 | 3

13. Secondary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) in Participants With Baseline Body Mass Index (BMI) ≥27 kg/m^2 at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted for baseline HbA1c. HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication were excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication, who had a BMI ≥27 kg/m^2 at baseline, and who had nonmissing HbA1c values at Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 113 | 118 | 109 | 104
Percent | -0.31 (0.0792) | -0.69 (0.0774) | -0.71 (0.0806) | -0.88 (0.0826)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.38, Standard Error of Mean 0.1109
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p = 0.0004, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -0.40, Standard Error of Mean 0.1129
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -0.57, Standard Error of Mean 0.1146

14. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose at Week 1 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Data after rescue medication was excluded from this analysis. Fasting plasma glucose was measured by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 1
Population: All randomized participants who received study medication and who had nonmissing fasting plasma glucose values at baseline and Week 1 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 126 | 120 | 121 | 115
mg/dL | 1.2 (1.934) | -6.0 (1.981) | -12.0 (1.976) | -16.5 (2.030)
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -7.1, Standard Error of Mean 2.769
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -13.1, Standard Error of Mean 2.762
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -17.7, Standard Error of Mean 2.808

15. Secondary Outcome: Adjusted Percentage of Participants Achieving Hemoglobin A1c (HbA1C) ≤6.5% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Percent adjusted for baseline HbA1c. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and who had HbA1c values at Baseline and Week 24 (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Number analyzed (Participants) | 18 | 29 | 18 | 36
Percentage of participants | 13.8 | 20.7 | 14.5 | 25.2
Statistical Analysis 1: Comparison: Placebo + Metformin vs Dapagliflozin, 2.5 mg + Metformin; Test type: Superiority or Other; Modified logistic regression — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 6.9
Statistical Analysis 2: Comparison: Placebo + Metformin vs Dapagliflozin, 5 mg + Metformin; Test type: Superiority or Other; p = 0.8627, Modified logistic regression; Mean Difference (Final Values) = 0.7
Statistical Analysis 3: Comparison: Placebo + Metformin vs Dapagliflozin, 10 mg + Metformin; Test type: Superiority or Other; p = 0.0149, Modified logistic regression — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = 11.3

ADVERSE EVENTS:
Groups:
- Dapagliflozin, 5.0 mg + Metformin: Participants received dapagliflozin, 5.0 mg, once daily plus open-label metformin ≥1500 mg per day for up to 102 weeks
Arm/Group | Placebo + Metformin | Dapagliflozin, 2.5 mg + Metformin | Dapagliflozin, 5.0 mg + Metformin | Dapagliflozin, 10 mg + Metformin
Serious Adverse Events (participants affected / at risk) | 14/137 | 15/137 | 9/137 | 14/135
Other Adverse Events (participants affected / at risk) | 84/137 | 87/137 | 77/137 | 83/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin (N=137) | Dapagliflozin, 2.5 mg + Metformin (N=137) | Dapagliflozin, 5.0 mg + Metformin (N=137) | Dapagliflozin, 10 mg + Metformin (N=135)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Necrobiosis (General disorders) | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin (N=137) | Dapagliflozin, 2.5 mg + Metformin (N=137) | Dapagliflozin, 5.0 mg + Metformin (N=137) | Dapagliflozin, 10 mg + Metformin (N=135)
Headache (Nervous system disorders) | 8 | 10 | 13 | 15
Hypertension (Vascular disorders) | 13 | 11 | 8 | 7
Influenza (Infections and infestations) | 15 | 19 | 20 | 17
Vomiting (Gastrointestinal disorders) | 2 | 6 | 7 | 4
Bronchitis (Infections and infestations) | 4 | 6 | 5 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 10 | 7 | 9 | 16
Dizziness (Nervous system disorders) | 7 | 5 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 7 | 18
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 5 | 5 | 7
Gastroenteritis (Infections and infestations) | 7 | 5 | 7 | 4
Nasopharyngitis (Infections and infestations) | 12 | 16 | 8 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 9 | 5 | 5
Urinary tract infection (Infections and infestations) | 8 | 5 | 8 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 10 | 4
Pharyngitis (Infections and infestations) | 3 | 7 | 5 | 8
Depression (Psychiatric disorders) | 2 | 8 | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 6 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.